CLINICAL TRIAL: NCT07031973
Title: The Effect of Micronutrient Supplementation in Combination With Healthy Lifestyle Coaching on Nutrition Status and Well-being: A 6-Month Intervention Study in Ghana
Brief Title: The Effect of Micronutrient Supplementation on Nutrition Status and Well-being
Acronym: NEXUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InnoNext Sarl (Industry)
Collaborators: University of Health and Allied Sciences (Other); HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PACTR202402872415588; UHAS-REC L.7 16123-24 (Other: UHAS RESEARCH ETHICAL COMMITTEE (REC))
Record Dates: First submitted 2025-02-15; First posted 2025-06-22 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Micronutrient Deficiencies
Keywords: Micronutrient deficiencies; Hidden Hunger; Sub-Saharan Africa

STUDY DESIGN:
Intervention Model Description: 1. Arm 1 will receive the daily Investigational Product (it will not be disclosed to the study participant if they receive a micronutrient supplement or a placebo) together with regular Nutrition Training and Healthy Lifestyle coaching
  2. Arm 2 will receive the daily micronutrient supplementation
  3. Arm 3 will receive the daily placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Arm 1: single blinded (Study participants unaware if active or placebo Investigational Product) Arm 2: double blinded Arm 3: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training and Active Ingredient Arm (Arm 1) (Active Comparator): Particiants receive a daily Investigational Product for 24 weeks plus Nutrition Training and Healthy Lifestyle Coaching
  Interventions: Dietary Supplement: Active Effervescent Powder; Other: Nutrition training and healthy lifestyle coaching
- Active Ingredient Arm (Arm 2) (Active Comparator): Participants receive a daily active Investigational Product for 24 weeks
  Interventions: Dietary Supplement: Active Effervescent Powder
- Placebo Arm (Arm 3) (Placebo Comparator): Participants receive a daily placebo Investigational Product for 24 weeks
  Interventions: Dietary Supplement: Placebo Effervescent powder

INTERVENTIONS:
Dietary Supplement: Active Effervescent Powder — Participants receive a daily sachet of effervescent powder that is Orange flavored, containing multiple vitamins and minerals
  Arms: Active Ingredient Arm (Arm 2); Training and Active Ingredient Arm (Arm 1)
Dietary Supplement: Placebo Effervescent powder — Participants receive a daily sachet of effervescent powder that is Orange flavored containing no active ingredients
  Arms: Placebo Arm (Arm 3)
Other: Nutrition training and healthy lifestyle coaching — Participants receive Nutrition training and healthy lifestyle coaching
  Arms: Training and Active Ingredient Arm (Arm 1)

SUMMARY:
Inadequate micronutrient status poses a significant challenge in Sub-Saharan African countries, including Ghana, and affects various demographics. The aim of the intervention study is to assess nutritional status and well-being through micronutrient supplementation with or without the combination of nutrition training and healthy lifestyle coaching among young adults in Ghana.

The outcomes the study is assessing are:

PRIMARY OUTCOME:

The primary outcome of this study is to determine if micronutrient supplement improves the vitamin D status of the study participants with or without additional Nutrition Training and Healthy Lifestyle Coaching. Vitamin D status will be assessed as serum 25(OH) D in serum.

SECONDARY OUTCOMES:

The secondary objectives are to:

1. determine if the provision of micronutrient supplement with or without additional NuTHLiC improves participants serum levels of vitamin B12, serum zinc, serum magnesium, serum ferritin and red blood cell Hb.
2. Assess the effect of micronutrient supplement with or without additional NuTHLiC on participants lifestyle habits and overall well- being through targeted questionnaires.

TRIAL DESIGN: This study is a 3-arm blinded randomized placebo-controlled trial among 151 young adults

participants in Arm 1 receive a daily Investigational Product and attend nutrition training and healthy lifestyle coaching;

participants in Arm 2 will receive an active Investigational Product;

participants in Arm 3 will receive a placebo Investigational Product.

Main data collection, including blood sampling for nutritional status will take place at Baseline (Day 0), Midpoint (Month 3) and Endpoint (Month 6). In addition, all participants will fill in a digital diary.

DETAILED DESCRIPTION:
This study is a 6-month intervention study to assess the effect of micronutrient supplementation in combination with healthy lifestyle coaching on nutrition status and well-being will improve nutritional status with or without the combination of nutrition training and healthy lifestyle coaching among young adults in Ghana.

The test product is an Effervescent powder that is Orange flavored containing multiple vitamins and minerals, in a single serving, packaged within a multi-layer structure foil sachet. Participants will be required to mix Effervescent powder with water before consumption.

The placebo is also an Effervescent powder that is Orange flavored, but without active components, packaged within a multi-layer structure foil sachet. The placebo will be packaged in a manner that it looks and feels just like the micronutrient supplement with the only difference being the absence of the active ingredient in the micronutrient supplement.

The primary outcome of this study is to determine if micronutrient supplement improves the vitamin D status of the study participants with or without additional Nutrition Training and Healthy Lifestyle Coaching (herein referred to as NuTHLiC), Vitamin D status will be assessed as serum 25(OH) D in serum.

The secondary objectives are to:

1. determine if the provision of micronutrient supplement with or without additional NuTHLiC improves participants serum levels of vitamin B12, serum zinc, serum magnesium, serum ferritin and red blood cell Hb.
2. Assess the effect of micronutrient supplement with or without additional NuTHLiC on participants lifestyle habits and overall well-being through targeted questionnaires

After consenting, blood samples will be taken for biochemical analyses and the participants will also be assessed through standardized questionnaires in addition to vitals and anthropometric measurements.

The primary analysis will be intention-to-treat analysis. We fit a linear mixed effect model involving a random effect of participants within treatment groups and fixed effects of time and their interactions. The treatment effects will be shown as the mean difference (95% CI) in the change in serum 25(OH)D concentration between intervention and control groups. Model assumptions will be checked by inspecting the residual and quantile-quantile plot. Difference-in-difference (DID) will be used to determine the effect of each micronutrient supplement between the treatment (intervention) groups and the control (placebo) group. Sub-group analysis will also be used to contrast the factorial analysis.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy students in their second and third years of study at University of Health and Allied Sciences, Fred N. Binka School of Public Health
* Females and males aged 18 - 25 years
* Agree to remain in the study area for the 26-week period of the follow-up
* Gives written informed consent

For female participants with childbearing potential:

* No plan to get pregnant the next 7 months (Acceptance of the requirement to use a highly effective form of birth control (herein referred to as condom) effective from consenting until at least week 24 after the final intake of Investigational Product (Month 6 visit).

Exclusion Criteria:

* Individuals taking routine micronutrient supplements
* History of food allergies
* Sensitivity to micronutrient supplement consumption and to any compositions of the micronutrients
* For females of child-bearing potential: pregnant as per serum pregnancy testing, or planning to become pregnant.
* Taking medications that could interact with the micronutrient supplements. Key medications which deplete the absorption of micronutrients include acid-suppressing and antacids, antiepileptic drugs (anti-convulsants), antibiotics, hormone replacement therapy (estrogens), digoxin, anti-inflammatory/analgesics
* Interested persons with severe anaemia (hemoglobin less than 7g/dl), as identified in the screening phase, will not be enrolled in the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved Vitamin D status | From baseline to endpoint data collection, the time frame is 24 weeks
  It will be measured with biomarker sampling at baseline, midpoint and endpoint if micronutrient supplementation improves the vitamin D status of the study participants with or without additional Nutrition Training and Healthy Lifestyle Coaching. Thresholds for determining Vitamin D status are based on serum 25-hydroxyvitamin D levels.

SECONDARY OUTCOMES:
Number of participants with improved vitamin B12 status | Time Frame: From baseline to endpoint data collection, the time frame is 24 weeks
  It will be measured with biomarker sampling at baseline, midpoint and endpoint if micronutrient supplementation improves the status of Vitamin B12 of the study participants that will receive a micronutrient supplement with or without additional Nutrition Training and Healthy Lifestyle Coaching.
Number of participants with improved serum zinc status | From baseline to endpoint data collection, the time frame is 24 weeks
  It will be measured with biomarker sampling at baseline, midpoint and endpoint if micronutrient supplementation improves the status of serum zinc of the study participants that will receive a micronutrient supplement with or without additional Nutrition Training and Healthy Lifestyle Coaching.
Number of participants with improved serum magnesium status | Time Frame: From baseline to endpoint data collection, the time frame is 24 weeks
  It will be measured with biomarker sampling at baseline, midpoint and endpoint if micronutrient supplementation improves the status of serum magnesium of the study participants that will receive a micronutrient supplement with or without additional Nutrition Training and Healthy Lifestyle Coaching.
Number of participants with improved serum ferritin and red blood cell Haemoglobin status | Time Frame: From baseline to endpoint data collection, the time frame is 24 weeks
  It will be measured with biomarker sampling at baseline, midpoint and endpoint if micronutrient supplementation improves the status of serum ferritin and red blood cell haemoglobin of the study participants that will receive a micronutrient supplement with or without additional Nutrition Training and Healthy Lifestyle Coaching.
Number of participants reporting effectiveness of additional Nutrition Training and Healthy Lifestyle Coaching on their lifestyle habits and overall well-being | From baseline to endpoint data collection, the time frame is 24 weeks
  The effect of micronutrient supplementation with or without additional Nutrition Training and Healthy Lifestyle Coaching on participants' lifestyle habits and overall well- being will be measured through targeted questionnaires as per outcome 2. The following data collection tools are used: 1) Global physical activity questionnaire; 2) Lifestyles and Habits Questionnaire; 3) Depression Anxiety Stress Scale 21; 4) Short Item Form Survey; 5) Young Women Food Intake; 6) Food Insecurity Experience; 7) 7-day Dietary Habit Recall; 8) Non-alcoholic Sugar-Sweetened Beverage Intake; 9) Multidimensional Subjective Wellbeing (MSW); 10) Nutrition Training and Healthy Lifestyle questionnaire. Each questionnaire has a different scale. Each questionnaire will be evaluated separately...

CONTACTS AND LOCATIONS:
Overall Officials: Francis B. Prof. Zotor, PhD, Principal Investigator — University of Health and Allied Sciences, Fred N. Binka School of Public Health (FNBSPH), Ghana
Locations (1):
- University of Health and Allied Sciences, Fred N. Binka School of Public Health, Hohoe, Volta Region, Ghana

IPD SHARING:
Plan to Share IPD: No
A Data sharing agreement (but not a formal IDP plan) was signed giving access to other researchers for academic, non-commercial purposes. It stipulates:
  1. For the sole use of any and all academic, non-commercial research purposes, including communication and publication in scientific journals, the Sponsor grants the Chief Investigator and the Participating Institution a royalty-free, non-exclusive, worldwide, perpetual, non-transferable license to use all Data, suitably anonymized.
  2. The Chief Investigator, shall not and shall procure that the Participating Institutions shall not, give access to the Data to any commercial organisation other than the Sponsor and the Supporting Funder during the term of this Agreement and for a period of five years from the date of completion of the Study without the prior written consent of the Sponsor.
  3. The Sponsor and the Chief Investigator agree to inform in writing each other about all organisations to whom they grant access to the Data.